CLINICAL TRIAL: NCT00126373
Title: A Randomized Controlled Trial of Wellbutrin for Crohn's Disease
Brief Title: A Trial of Wellbutrin for Crohn's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Altschuler, Eric, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGO10410022
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Crohn Disease
Keywords: Crohn disease; TNF-alpha
MeSH Terms: conditions — Crohn Disease | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo (sugar) pill with identical look to bupropion
  Interventions: Drug: Wellbutrin (bupropion)
- buproprion (Experimental): bupropion pill
  Interventions: Drug: Wellbutrin (bupropion)

INTERVENTIONS:
Drug: Wellbutrin (bupropion) — bupropion 150mg-300mg daily
  Other Names: Wellbutrin, bupropion

SUMMARY:
The investigators are testing the hypothesis that Wellbutrin (bupropion) can give a clinical remission in Crohn's disease.

DETAILED DESCRIPTION:
Wellbutrin (bupropion) is approved for use as an antidepressant. There have been some cases in which people on Wellbutrin had significant improvement clinically in their Crohn's disease. In this trial, the hypothesis that Wellbutrin can induce clinical remission in Crohn's disease will be tested. The investigators will also be looking to see if Wellbutrin can lower levels of the inflammatory cytokine tumor necrosis factor-alpha (TNF).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Crohn's disease with 220 < CDAI < 400.
* All patients in the study must have not had any anti-TNF antibodies for at least eight weeks.

Exclusion Criteria:

* Patients will be excluded from the study if they have fulminant Crohn's disease requiring parenteral steroid treatment, hospitalization, or need of surgery imminently.
* Patients with serious infections in the preceding three months, opportunistic infections within one month, or current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurological, or cerebral disease will be excluded.
* Patients will also be excluded from the study if they have a history of a seizure, epilepsy, presumed current central nervous system tumor, have or have had anorexia nervosa or bulimia, are currently taking or have taken in the last four weeks any drug in the monoamine oxidase inhibitor class, or are allergic to Wellbutrin.
* Patients with active major depression or suicidal ideation will be excluded, as will patients with a score of 19 or higher on the Beck depression inventory.
* Patients will be excluded if they are currently or have taken a medicine in the selective serotonin reuptake class, mirtazapine, venlafaxine, a tricyclic antidepressant, a mood stabilizing, or antipsychotic medication in the previous two weeks.
* Patients will be excluded if they are currently abusing alcohol or have alcohol dependence.
* Patients will be excluded from the study if their baseline liver function tests are greater than twice the upper limit of normal, or if a clinical investigator believes that their baseline chemistry, liver function tests or complete blood count contraindicates entry into the study.
* Pregnant or lactating females are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with Crohn's disease activity index (CDAI) < 150 at the end of twelve weeks | 0, 2, 4, 8, 12 weeks

SECONDARY OUTCOMES:
Number of patients with CDAI drop of at least 70 points at the end of twelve weeks | 0, 12 weeks
Time course of CDAI | 0, 2, 4, 8, 12 weeks
Effect of drug and/or placebo on tumor necrosis factor-alpha (TNF) levels | 0, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Altschuler, M.D., Ph.D., Principal Investigator — Mt. Sinai Medical Center
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Mt. Sinai Medical Center, New York, New York